CLINICAL TRIAL: NCT01478477
Title: Prevention of Aromatase Inhibitor-Induced Joint Symptoms With Omega 3 Fatty Acid Supplementation: a Randomized Placebo Controlled Pilot Study
Brief Title: Omega-3 Fatty Acids in Preventing Joint Symptoms in Patients With Stage I-III Breast Cancer Receiving Anastrozole, Exemestane, or Letrozole
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Cancer and Leukemia Group B (Network)
Responsible Party: Principal Investigator, Nicole Williams, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OSU-11022; NCI-2011-03262 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-11-14; First posted 2011-11-23 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Recurrent Breast Cancer; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fish Oils; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm I (omega-3 fatty acid supplement) (Experimental): Omega 3 Polyunsaturated Fatty Acids(n-3 PUFA)
  Interventions: Dietary Supplement: omega-3 fatty acid supplement; Other: Clinical assessments; Other: Assessment of therapy complications; Procedure: Magnetic Resonance Imaging; Procedure: Correlative/special studies
- Arm II (placebo) (Placebo Comparator): Typical American Diet oils (TAD)
  Interventions: Other: Placebo; Other: Clinical assessments; Other: Assessment of therapy complications; Procedure: Magnetic Resonance Imaging; Procedure: Correlative/special studies
- Clinical Assessments (Experimental): Brief Pain Inventory (BPI), Stanford's Health Assessment-Disability Index (HAS), FACT-B and endocrine subscale (FACT-ES)
  Interventions: Dietary Supplement: omega-3 fatty acid supplement; Other: Placebo
- Assessment of therapy complications (Experimental): Adverse events will be monitored by self-reporting of signs and symptoms. Patients will maintain a daily diary of time of supplement intake and any possible ill effects, with instructions to contact the PI or Research Nurse to discuss and manage any possible side effects.
  Interventions: Dietary Supplement: omega-3 fatty acid supplement; Other: Placebo
- Magnetic Resonance Imaging (Experimental): Optional bilateral hand and wrist MRI imaging will be obtained
  Interventions: Dietary Supplement: omega-3 fatty acid supplement; Other: Placebo
- Correlative/special studies (Experimental): Enrolled participants will have peripheral blood samples drawn for plasma and RBC n-3 PUFA levels within 4 weeks of starting AI therapy.
  Interventions: Dietary Supplement: omega-3 fatty acid supplement; Other: Placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acid supplement — 6 capsules per day (4.3 g)x 6 months
  Other Names: fish oil; omega fatty acid; O3FA; MNSG-194®; n-3 PUFA supplementation
  Arms: Arm I (omega-3 fatty acid supplement); Assessment of therapy complications; Clinical Assessments; Correlative/special studies; Magnetic Resonance Imaging
Other: Placebo — 6 capsules per day (4.3 g)x 6 months. Supplement should be taken with food once per day. No specific food requirements are needed.
  Other Names: PLCB; Typical American Diet oils; TAD
  Arms: Arm II (placebo); Assessment of therapy complications; Clinical Assessments; Correlative/special studies; Magnetic Resonance Imaging
Other: Clinical assessments — All three instruments will be administered at baseline, at 3 months, 6 months and at additional time intervals when there is a significant change in therapy (discontinuation/switch, pain medication administration) during routine medical oncology visits.
  Other Names: Brief Pain Inventory; BPI; Stanford's Health Assessment-Disability Index; HAS; FACT-B and endocrine subscale; FACT-ES
  Arms: Arm I (omega-3 fatty acid supplement); Arm II (placebo)
Other: Assessment of therapy complications — Severity/grade of reaction according to the NCI Common Terminology Criteria for Adverse Events v4.0 (CTCAE).
  Other Names: adverse events; toxicities; Expected Toxicities; Potential Toxicities
  Arms: Arm I (omega-3 fatty acid supplement); Arm II (placebo)
Procedure: Magnetic Resonance Imaging — Optional bilateral hand and wrist MRI imaging will be obtained at baseline and at 6 months to eligible patients who have no contraindications to MRI imaging.
  Other Names: MRI; NMR imaging; NMRI; nuclear magnetic resonance imaging
  Arms: Arm I (omega-3 fatty acid supplement); Arm II (placebo)
Procedure: Correlative/special studies — Plasma, RBC, and serum samples from the baseline blood draw will also be stored at -70C for fatty acid and biomarker analyses and repeated at 3 month and 6 month intervals. Samples will be analyzed in batches every 6 months.
  Other Names: laboratory studies
  Arms: Arm I (omega-3 fatty acid supplement); Arm II (placebo)

SUMMARY:
This randomized pilot trial studies omega-3 fatty acid in preventing joint symptoms in patients with stage I-III breast cancer receiving anastrozole, exemestane, or letrozole. Omega-3 fatty acid supplement may lessen or prevent joint stiffness or pain in patients receiving hormone therapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess the feasibility of evaluating joint symptoms in postmenopausal women with breast cancer randomized to n-3 PUFA (omega-3 fatty acid) vs. placebo supplementation using the Functional Assessment of Cancer Therapy-Breast (FACT-B) and endocrine subscale (FACT-ES), Brief Pain Inventory (BPI) and Stanford's Health Assessment -Disability Index (HAS) during the first 6 months of adjuvant aromatase inhibitor (AI) therapy.

II. To preliminarily evaluate the efficacy of n-3 PUFA vs. placebo supplementation on AI induced joint symptoms.

III. To explore blood and imaging based biomarkers (plasma and red blood cell [RBC] levels of n-3 PUFAs, inflammatory cytokines and receptors, and intra-articular tenosynovial inflammation by musculoskeletal magnetic resonance imaging [MRI] imaging) of AI-induced joint symptoms in women on AI therapy randomized to n-3 PUFAs vs. placebo supplementation.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive omega-3 fatty acid orally (PO) once daily (QD) for 6 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO QD for 6 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer stages I-III initiating first adjuvant AI therapy with any of the Food and Drug Administration- (FDA) approved AIs (anastrozole, exemestane, letrozole)
* Concurrent gonadotropin-releasing hormone (GnRH) agonist therapy is allowed
* Concurrent breast related radiation therapy is allowed
* Prior tamoxifen use is allowed
* Prior chemotherapy is allowed
* History of osteoarthritis and/or fibromyalgia is allowed
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Metastatic malignancy of any kind
* Rheumatoid arthritis and other types of autoimmune and inflammatory joint disease, with the exception of osteoarthritis and fibromyalgia
* AI use > 2 weeks prior to study enrollment
* Known bleeding disorders
* History of diabetes mellitus, heart disease or TIA/stroke
* Current use of warfarin or other anticoagulants
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia,or psychiatric illness/social situation that would limit compliance with study requirements
* Daily use of n-3 PUFA concentrates or capsules or regular or any other supplements that might interact with n-3 PUFA supplements within six months of study initiation; sporadic use of n-3 PUFA supplement may be eligible if there has been a 3-month washout period prior to randomization
* Pregnant or nursing women
* Known sensitivity or allergy to fish or fish oil
* Concurrent use of daily full dose aspirin (≥ 325 mg/day), nonsteroidal anti-inflammatory drugs (NSAIDs) or NSAID-containing products or steroids; one month washout period is required prior to randomization
* Unable to give informed consent
* In patients consenting for optional MRIs, any contraindication to MRI examination including but not limited to ferromagnetic metal in the body, pacemaker, or severe claustrophobia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-10-04 (Actual); Primary Completion 2014-01-09 (Actual); Study Completion 2014-01-09 (Actual)

PRIMARY OUTCOMES:
Pain score change after 6 months (6 months -baseline) based on the FACT-B/ES instrument | baseline, 6 months
  Pain scores based on FACT-B/ES, HAS and BPI will be plotted over time for each arm. Agreement between HAS, BPI-short and FACT-B/ES evaluated using Altman and Bland plot after proper data transformation. Also, Linear Mixed model used to explore if the pain scores are different at 3 and 6 months. Logistic regression models used to compare the occurrence of moderate to severe joint symptoms during the 6 month period between the two treatment groups, with potential covariates including age, body mass index, baseline pain scores (0 month), prior chemotherapy and other variables.

SECONDARY OUTCOMES:
Pain score change after 6 months (6 months -baseline) based on the HAS and BPI instruments | baseline, 6 months
  Agreement between HAS, BPI-short and FACT-B/ES evaluated using Altman and Bland plot after proper data transformation. Also, Linear Mixed model used to explore if the pain scores are different at 3 and 6 months. Logistic regression models used to compare the occurrence of moderate to severe joint symptoms during the 6 month period between the two treatment groups, with potential covariates including age, body mass index, baseline pain scores (0 month), prior chemotherapy and other variables.
Compliance rates with oral supplements (omega-3 fatty acid and placebo) | baseline, 6 months
Feasibility of using the instruments HAS, BPI-short, FACT-B/ES for the assessment of joint symptoms | baseline, 6 months
Effectiveness of blinding | baseline, 6 months
  Summarized using a Chi-square test.
Correlation of guess with pain scores | baseline, 6 months
  Checked using logistic models to see if treatment guesses are explained by the patient's awareness of clinical benefit.
Relationship between serum and RBC omega-3 fatty acid levels, inflammatory blood markers and MRI changes and the joint symptoms | baseline, 6 months
  Scatter plots and correlation coefficients (either Pearson or Spearman) will be used to summarize their pair wise relation. The differences between the treatment and placebo in terms of these measures will also be reported using numerical summaries and graphic plots.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Williams, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Orchard TS, Andridge RR, Yee LD, Lustberg MB. Diet Quality, Inflammation, and Quality of Life in Breast Cancer Survivors: A Cross-Sectional Analysis of Pilot Study Data. J Acad Nutr Diet. 2018 Apr;118(4):578-588.e1. doi: 10.1016/j.jand.2017.09.024. Epub 2017 Dec 9. PMID 29233615
- See also: Jamesline — http://cancer.osu.edu